CLINICAL TRIAL: NCT01871194
Title: An Observational Post-Authorization Safety Specialist Cohort Event Monitoring Study (SCEM) to Monitor the Safety and Utilization of Rivaroxaban (Xarelto®) for the Prevention of Stroke in Patients With Atrial Fibrillation (AF), Treatment of Deep Vein Thrombosis (DVT) and Pulmonary Embolism (PE), and the Prevention of Recurrent DVT and PE in the Secondary Care Hospital Setting in England and Wales.
Brief Title: An Observational Post-Authorization Safety Specialist Cohort Event Monitoring Study (SCEM) to Monitor the Safety and Utilization of Rivaroxaban (Xarelto®).
Acronym: ROSE
Status: Completed | Type: Observational
Sponsor: Professor Saad Shakir (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor-Investigator, Professor Saad Shakir, Director, Drug Safety Research Unit, Southampton, UK
Organization: Drug Safety Research Unit, Southampton, UK (Other)
Other Study IDs: ROSE
Record Dates: First submitted 2013-05-29; First posted 2013-06-06 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Atrial Fibrillation; Deep Vein Thrombosis; Pulmonary Embolism
MeSH Terms: conditions — Atrial Fibrillation; Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Rivaroxaban: This is a non-interventional study
- Alternative anticoagulant therapy: This is a non-interventional study

SUMMARY:
This study aims to evaluate the use of rivaroxaban and its short term safety when used by patients for the new indications of prevention of stroke and systemic embolism in patients with non-valvular atrial fibrillation, treatment of deep vein thrombosis (DVT) and pulmonary embolism (PE) and prevention of recurrent DVT and PE. Any adult patient started by their care team on rivaroxaban or an alternative anticoagulant for the specified indications during the study period will be eligible to take part. A questionnaire will be completed by the care team of each patient at the start of treatment and again 12 weeks later. The care team will complete the questionnaires using information from the patient's medical notes, not by asking the patient directly. If a participant has an adverse event during the 12 week period, we may ask the patient's care team to fill out a further follow up questionnaire. No other examinations or tests will be performed. Patients will only be recruited to the study after the clinical decision to prescribe rivaroxaban or an alternative anticoagulant has been made, so that prescribing behaviour is not altered by the study. It is an observational, non-interventional study covering the whole of England and Wales.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or above after study start
* index date on or after study start
* signed, informed consent
* patients treated for DVT or PE
* patients with non-valvular AF (with one or more risk factors) treated for prevention of stroke and systemic embolism

Exclusion Criteria:

* any use of univalent direct thrombin inhibitor or direct factor Xa inhibitors
* use of anticoagulant therapy or other vitamin K antagonists recorded within one year prior to index date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients prescribed rivaroxaban or an alternative anticoagulant in the secondary care hospital setting in England and Wales for the prevention of stroke in patients with AF, the treatment of DVT or PE, or the prevention of recurrent DVT and PE.
Sampling Method: Non-Probability Sample
Enrollment: 3400 (Actual)
Dates: Start 2013-05; Primary Completion 2016-01 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Cumulative incident risk of haemorrhage within gastrointestinal and urogenital organ sites (which meets the criteria for a major bleed) and all intracranial sites. | During 12 weeks after initiation of treatment with rivaroxaban or alternative anticoagulant therapy
  The cumulative incidence will be calculated according to the formula:
  Total number of new cases during 12 week observation period x 100 / Population initially at risk
  If the observed cumulative incidence from this study falls within the range expected as set by the precision limits of cumulative incidence from clinical trial data, then the null hypothesis (of no difference) will not be rejected.

CONTACTS AND LOCATIONS:
Locations (1):
- Drug Safety Research Unit, Southampton, Hampshire, United Kingdom

REFERENCES:
- [Derived] Evans A, Davies M, Osborne V, Roy D, Shakir S. Evaluation of the incidence of bleeding in patients prescribed rivaroxaban for the treatment and prevention of deep vein thrombosis and pulmonary embolism in UK secondary care: an observational cohort study. BMJ Open. 2020 Nov 3;10(11):e038102. doi: 10.1136/bmjopen-2020-038102. PMID 33148732